CLINICAL TRIAL: NCT07021664
Title: Santé, Imagerie et Cognition à Travers la Transition ménopausique
Brief Title: Health, Imaging, and Cognition Across the Menopausal Transition
Acronym: MOSAIC
Status: Not yet recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Nestlé Health Science (Industry)
Responsible Party: Sponsor
Other Study IDs: 2025-58-28
Record Dates: First submitted 2025-04-24; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Menopause
Keywords: menopause; cognition; metabolism; estrogen; ketone; PET scan; estrogen receptor
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood and plasma will be retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- premenopause: Women between 35 and 55 years old who still have regular menstrual cycles, with no noticeable changes in the past 10 months.
- perimenopause: Women between 40 and 60 years old who have experienced changes in their menstrual cycles, such as irregular timing (varying by more than 7 days) for at least 10 cycles, or no period for 3 to 11 months.
- postmenopause: Women between 45 and 65 years old who have not had a menstrual period for 12 months or more.

SUMMARY:
This observational cross-sectional study aims to better understand how the menopausal transition affects brain energy metabolism and cognition. Menopause, a natural stage in a woman's life, is typically divided into three phases: premenopause, perimenopause, and postmenopause. This transition involves hormonal fluctuations and a decline in estrogen levels, which can impact physical, emotional, and cognitive well-being. Common symptoms include hot flashes, sleep disturbances, mood changes, and difficulties with memory and concentration.

Emerging evidence suggests that the decline in estrogen may impair how the brain uses glucose, its primary energy source. This reduction in glucose metabolism is thought to contribute to cognitive difficulties reported during midlife. In contrast, the brain's capacity to use ketones-alternative energy substrates produced during fasting or low-carbohydrate intake-appears preserved during aging and hormonal changes. Increasing circulating ketones may offer a promising strategy to support brain energy and cognitive function.

To explore these relationships, the study will employ advanced brain imaging (PET scans) to assess glucose and ketone uptake in the brain. Additional measures will include hormone levels, cognitive testing, continuous glucose monitoring, and MRI. PET tracers will also be used to evaluate estrogen receptor distribution, providing insight into how the brain responds to hormonal changes.

A total of 45 women aged 35-60 will be enrolled and categorized into three groups (15 per group): premenopause, perimenopause, and postmenopause. Each participant will attend four study visits that include questionnaires, blood tests, cognitive assessments, metabolic measurements, and imaging procedures.

The results may help identify early neurobiological and metabolic markers associated with the menopausal transition. These findings could inform new approaches to preserve brain health and prevent cognitive decline in aging women. Improving understanding of how the female brain adapts to hormonal shifts may ultimately support more targeted strategies for promoting healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and speak French
* Capable of understanding and signing informed consent GROUP SPECIFIC INCLUSION CRITERIA Premenopause: • Women aged 35 to 55; No change in menstrual cycle regularity over the past 10 months (variation less than 7 days per cycle)

Perimenopause: Women aged 40 to 60; Menstrual cycles varying by more than 7 days per cycle for at least 10 cycles, or no period for 3 to 11 months

postmenopause: Women aged 45 to 65; No menstrual period for ≥ 12 months

Exclusion Criteria:

* Pregnancy, childbirth within the past 12 months, or breastfeeding
* Use of hormone replacement therapy or hormonal contraceptives in the past 6 months
* contraindications to MRI (e.g., presence of non-compatible metallic objects)
* Claustrophobia
* Type 1 diabetes
* Adherence to a ketogenic intervention (e.g., ketone supplements, intermittent fasting, ketogenic diet) in the past 3 months
* Engaging in intense physical activity 5 times per week or more
* Any significant neurological disorder (e.g., dementia, brain tumor, seizure disorder, history of significant head trauma with persistent neurological deficits, known structural brain abnormalities)
* History of oophorectomy or hysterectomy
* Any significant psychiatric disorder (e.g., major depression within the past 2 years, bipolar disorder, schizophrenia)
* Systemic diseases or unstable/uncontrolled medical conditions (e.g., cardiovascular disease, uncontrolled diabetes, kidney or liver disorders)
* Any other condition that may interfere with participation, as judged by the study physician

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy individuals from the general population
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
cerebral metabolic rates (μmol/100 g/min) measured by PET (11C-AcAc +18F-FDG) | 1 day at baseline
  Brain energy metabolism will be quantified using two PET tracers: 11C-acetoacetate (for ketone use) and 18F-fluorodeoxyglucose (for glucose use). This will allow comparison of brain fuel usage between three menopausal groups (PRE, PERI, POST).Total Cerebral metabolic rates (μmol/100 g/min) (CMR tot= CMR acac + CMRglu)
Tracer influx rates (k) measured by PET (11C-AcAc +18F-FDG) | 1 day at baseline
  Brain energy metabolism will be quantified using two PET tracers: 11C-acetoacetate (for ketone use) and 18F-fluorodeoxyglucose (for glucose use). This will allow comparison of brain fuel usage between three menopausal groups (PRE, PERI, POST). tracer influx rates (K values).

SECONDARY OUTCOMES:
Time-activity curves of the estrogen receptor in the brain (by 18F-4FMFES PET) | 1 day at baseline
  Time-activity curves of the estrogen recept will be measured using 18F-4FMFES PET express as SUV (Standardized Uptake Value)
distribution volume ratio of the estrogen receptor in the brain (by 18F-4FMFES PET) | 1 day at baseline
  distribution volume ratio of the estrogen receptor will be measured by kinetic modelisation using 18F-4FMFES PET.
Glucose variability (SD of glucose measured by continuous glucose monitoring) | Over 5 days following sensor placement et stabilisation
  Continuous glucose monitoring (CGM) will track glucose levels over several days. Glycemic variability will be assessed by the standard deviation of glucose values over the 5 days monitoring period. (mmol/L)
Glucose average (mean of glucose measured by continuous glucose monitoring) | Over 5 days following sensor placement et stabilisation
  Continuous glucose monitoring (CGM) will track glucose levels over several days. Average glucose concentration over the monitoring period.(mmol/L)
Time in range | Over 5 days following sensor placement et stabilisation
  Total minutes with glucose values within the standard glycemic range (3.9-10.0 mmol/L) over the 5 days monitoring period. (min)

OTHER OUTCOMES:
Brain volume | 1 day at baseline
  Will be measured by MRI - T1-weighted images and express in cm³
Rey Auditory Verbal Learning Test (RAVLT) | 1 day at baseline
  Assesses verbal memory. Total score (range: 0-75); higher scores indicate better performance
Stroop Color and Word test (Stroop Test) (secondes) | 1 day at baseline
  Measures processing speed and executive function; outcome is time to completion.
  Unit of Measure: Seconds; lower scores indicate better performance
Trail making test (secondes) | 1 day at baseline
  Assesses cognitive flexibility, visual attention, and processing speed. Unit of Measure: Seconds; lower scores indicate better performance
Montreal Cognitive Assessment (MoCA) score | 1 day at baseline
  Global cognitive screening tool. Unit of Measure: Score (range: 0-30); higher scores indicate better cognition.
Boston naming tests (total answer) | 1 day at baseline
  Measures language and word retrieval ability.Total correct responses (range: 0-60); higher scores are better
Symbol coding (score) | 1 day at baseline
  Assesses processing speed.Score (higher = better)
Logical Memory Subtest of the Wechsler Memory Scale-IV | 1 day at baseline
  Assesses elayed story recall. Score (0-25); higher scores indicate better memory
Fasting plasma glucose (mM) | 1 day at baseline
  Blood samples will be used to assess the systemic metabolis plasma markers and will be compared across 3 groups
Fasting plasma insulin (mM) | 1 day at baseline
  Blood samples will be used to assess the systemic metabolis plasma markers and will be compared across 3 groups
Fasting plasma HbA1c (%) | 1 day at baseline
  Blood samples will be used to assess the systemic metabolis plasma markers and will be compared across 3 groups
Fasting plasma total ketone (uM) | 1 day at baseline
  Blood samples will be used to assess the systemic metabolis plasma markers and will be compared across 3 groups. Total ketone = acetoacetate + beta-hydroxybutyrate
Estrogene levels (pmol/L) | 1 day at baseline
  Blood samples will be used to assess sex hormone and will be compared across 3 group
follicule stimulating hormone levels (mIU/mL) | 1 day at baseline
  Blood samples will be used to assess sex hormone and will be compared across 3 group
Progesterone (nmol/L) | 1 day at baseline
  Blood samples will be used to assess sex hormone and will be compared across 3 group
hormone lutéinisante (mUI/mL) | 1 day at baseline
  Blood samples will be used to assess sex hormone and will be compared across 3 group
Menopause-Specific Quality of Life Questionnaire | 1 day at baseline
  Self-reported questionnaires. Self-reported symptom burden. Unit of Measure: Score (range: 0-44); higher = more severe symptoms
Menopause Rating Scale | 1 day at baseline
  Self-reported symptom burden. Unit of Measure: Score (range: 0-44); higher = more severe symptoms
Pittsburgh Sleep Quality Index | 1 day at baseline
  Self-reported questionnaire. Assesses sleep quality over the past month. Unit of Measure: Score (range: 0-21); higher = poorer sleep
Patient Health Questionnaire (PHQ-9) | 1 day at baseline
  Depressive symptoms. Score (range: 0-27); higher = more severe depression
Subjective memory complain | 1 day at baseline
  Self-reported memory or concentration issues. Unit of Measure: Score (range 62-372) ; higher scores indicate more complaints
International Physical Activity Questionnaire | 1 day at baseline
  Physical activity over the past week. (MET-minutes/week)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, Ph.D, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le Vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
There is no current plan to share individual participant data (IPD) with external researchers. While data reuse within the study team is permitted, external data sharing is subject to sponsor agreement and may be considered on a case-by-case basis in the future.

REFERENCES:
- [Background] Andy C, Nerattini M, Jett S, Carlton C, Zarate C, Boneu C, Fauci F, Ajila T, Battista M, Pahlajani S, Christos P, Fink ME, Williams S, Brinton RD, Mosconi L. Systematic review and meta-analysis of the effects of menopause hormone therapy on cognition. Front Endocrinol (Lausanne). 2024 Mar 4;15:1350318. doi: 10.3389/fendo.2024.1350318. eCollection 2024. PMID 38501109
- [Background] Castellano CA, Baillargeon JP, Nugent S, Tremblay S, Fortier M, Imbeault H, Duval J, Cunnane SC. Regional Brain Glucose Hypometabolism in Young Women with Polycystic Ovary Syndrome: Possible Link to Mild Insulin Resistance. PLoS One. 2015 Dec 9;10(12):e0144116. doi: 10.1371/journal.pone.0144116. eCollection 2015. PMID 26650926
- [Background] Mosconi L, Nerattini M, Matthews DC, Jett S, Andy C, Williams S, Yepez CB, Zarate C, Carlton C, Fauci F, Ajila T, Pahlajani S, Andrews R, Pupi A, Ballon D, Kelly J, Osborne JR, Nehmeh S, Fink M, Berti V, Dyke JP, Brinton RD. In vivo brain estrogen receptor density by neuroendocrine aging and relationships with cognition and symptomatology. Sci Rep. 2024 Jun 20;14(1):12680. doi: 10.1038/s41598-024-62820-7. PMID 38902275
- [Background] Paquette M, Phoenix S, Lavallee E, Rousseau JA, Guerin B, Turcotte EE, Lecomte R. Cross-Species Physiological Assessment of Brain Estrogen Receptor Expression Using 18F-FES and 18F-4FMFES PET Imaging. Mol Imaging Biol. 2020 Oct;22(5):1403-1413. doi: 10.1007/s11307-020-01520-w. Epub 2020 Jul 22. PMID 32699974
- [Background] Arjmand S, Bender D, Jakobsen S, Wegener G, Landau AM. Peering into the Brain's Estrogen Receptors: PET Tracers for Visualization of Nuclear and Extranuclear Estrogen Receptors in Brain Disorders. Biomolecules. 2023 Sep 18;13(9):1405. doi: 10.3390/biom13091405. PMID 37759805
- [Background] Fortier M, Castellano CA, St-Pierre V, Myette-Cote E, Langlois F, Roy M, Morin MC, Bocti C, Fulop T, Godin JP, Delannoy C, Cuenoud B, Cunnane SC. A ketogenic drink improves cognition in mild cognitive impairment: Results of a 6-month RCT. Alzheimers Dement. 2021 Mar;17(3):543-552. doi: 10.1002/alz.12206. Epub 2020 Oct 26. PMID 33103819
- [Background] Fortier M, Castellano CA, Croteau E, Langlois F, Bocti C, St-Pierre V, Vandenberghe C, Bernier M, Roy M, Descoteaux M, Whittingstall K, Lepage M, Turcotte EE, Fulop T, Cunnane SC. A ketogenic drink improves brain energy and some measures of cognition in mild cognitive impairment. Alzheimers Dement. 2019 May;15(5):625-634. doi: 10.1016/j.jalz.2018.12.017. Epub 2019 Apr 23. PMID 31027873
- [Background] Croteau E, Castellano CA, Richard MA, Fortier M, Nugent S, Lepage M, Duchesne S, Whittingstall K, Turcotte EE, Bocti C, Fulop T, Cunnane SC. Ketogenic Medium Chain Triglycerides Increase Brain Energy Metabolism in Alzheimer's Disease. J Alzheimers Dis. 2018;64(2):551-561. doi: 10.3233/JAD-180202. PMID 29914035
- [Background] Cunnane SC, Trushina E, Morland C, Prigione A, Casadesus G, Andrews ZB, Beal MF, Bergersen LH, Brinton RD, de la Monte S, Eckert A, Harvey J, Jeggo R, Jhamandas JH, Kann O, la Cour CM, Martin WF, Mithieux G, Moreira PI, Murphy MP, Nave KA, Nuriel T, Oliet SHR, Saudou F, Mattson MP, Swerdlow RH, Millan MJ. Brain energy rescue: an emerging therapeutic concept for neurodegenerative disorders of ageing. Nat Rev Drug Discov. 2020 Sep;19(9):609-633. doi: 10.1038/s41573-020-0072-x. Epub 2020 Jul 24. PMID 32709961
- [Background] Mosconi L, Brinton RD. How would we combat menopause as an Alzheimer's risk factor? Expert Rev Neurother. 2018 Sep;18(9):689-691. doi: 10.1080/14737175.2018.1510320. Epub 2018 Aug 13. No abstract available. PMID 30091648
- [Background] Mosconi L, Berti V, Quinn C, McHugh P, Petrongolo G, Osorio RS, Connaughty C, Pupi A, Vallabhajosula S, Isaacson RS, de Leon MJ, Swerdlow RH, Brinton RD. Perimenopause and emergence of an Alzheimer's bioenergetic phenotype in brain and periphery. PLoS One. 2017 Oct 10;12(10):e0185926. doi: 10.1371/journal.pone.0185926. eCollection 2017. PMID 29016679
- [Background] Mosconi L, Berti V, Quinn C, McHugh P, Petrongolo G, Varsavsky I, Osorio RS, Pupi A, Vallabhajosula S, Isaacson RS, de Leon MJ, Brinton RD. Sex differences in Alzheimer risk: Brain imaging of endocrine vs chronologic aging. Neurology. 2017 Sep 26;89(13):1382-1390. doi: 10.1212/WNL.0000000000004425. Epub 2017 Aug 30. PMID 28855400
- [Background] Snyder HM, Asthana S, Bain L, Brinton R, Craft S, Dubal DB, Espeland MA, Gatz M, Mielke MM, Raber J, Rapp PR, Yaffe K, Carrillo MC. Sex biology contributions to vulnerability to Alzheimer's disease: A think tank convened by the Women's Alzheimer's Research Initiative. Alzheimers Dement. 2016 Nov;12(11):1186-1196. doi: 10.1016/j.jalz.2016.08.004. Epub 2016 Sep 27. PMID 27692800
- [Background] Gold EB, Sternfeld B, Kelsey JL, Brown C, Mouton C, Reame N, Salamone L, Stellato R. Relation of demographic and lifestyle factors to symptoms in a multi-racial/ethnic population of women 40-55 years of age. Am J Epidemiol. 2000 Sep 1;152(5):463-73. doi: 10.1093/aje/152.5.463. PMID 10981461
- [Background] Delanerolle G, Phiri P, Elneil S, Talaulikar V, Eleje GU, Kareem R, Shetty A, Saraswath L, Kurmi O, Benetti-Pinto CL, Muhammad I, Rathnayake N, Toh TH, Aggarwal IM, Shi JQ, Taylor J, Riach K, Potocnik K, Litchfield I, Kemp HF, Briggs P; MARIE collaborative. Menopause: a global health and wellbeing issue that needs urgent attention. Lancet Glob Health. 2025 Feb;13(2):e196-e198. doi: 10.1016/S2214-109X(24)00528-X. Epub 2024 Dec 18. No abstract available. PMID 39708829
- [Background] Harlow SD, Gass M, Hall JE, Lobo R, Maki P, Rebar RW, Sherman S, Sluss PM, de Villiers TJ; STRAW + 10 Collaborative Group. Executive summary of the Stages of Reproductive Aging Workshop + 10: addressing the unfinished agenda of staging reproductive aging. J Clin Endocrinol Metab. 2012 Apr;97(4):1159-68. doi: 10.1210/jc.2011-3362. Epub 2012 Feb 16. PMID 22344196
- [Background] Mosconi L, Rahman A, Diaz I, Wu X, Scheyer O, Hristov HW, Vallabhajosula S, Isaacson RS, de Leon MJ, Brinton RD. Increased Alzheimer's risk during the menopause transition: A 3-year longitudinal brain imaging study. PLoS One. 2018 Dec 12;13(12):e0207885. doi: 10.1371/journal.pone.0207885. eCollection 2018. PMID 30540774